CLINICAL TRIAL: NCT05936255
Title: Pilot Examination of a Telehealth, Cognitive-behavioral Therapy for Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low feasibility of participant recruitment.
Sponsor: Florida State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Victor Buitron, Principal Investigator, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003755; U54CA267730 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Suicide Prevention; Suicidal Ideation
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Give to Others Module (Experimental): A brief, talk therapy protocol that targets negative interpersonal beliefs (i.e., perceived social disconnection, burdensomeness) using cognitive-behavioral strategies.
  Interventions: Behavioral: Give to Others Module

INTERVENTIONS:
Behavioral: Give to Others Module — Negative interpersonal beliefs are targeted via cognitive-behavioral strategies, including evaluation of cognitive distortions, and activity planning and tracking.

SUMMARY:
This project is designed to refine a 6-week telehealth therapy intervention targeting negative interpersonal beliefs among community-dwelling youth with elevated levels of psychopathology. The study design is a single-arm open trial. The intervention is comprised of weekly teen and parent group cognitive-behavioral therapy, regular check-ins with the youths, and a module embedded throughout treatment that targets negative interpersonal beliefs (i.e., perceived social disconnection, burdensomeness). The goal of the study is to evaluate the feasibility of the treatment and assessment protocol, refine the intervention based on qualitative feedback, and evaluate changes in negative interpersonal beliefs. Youths complete two qualitative interviews about their interpersonal relationships and their feedback about the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years of age
* endorsement of perceived burdensomeness (score of greater than 3 on the Interpersonal Needs Questionnaire)
* emotional/behavioral problems broadly defined (Pediatric Symptom Checklist score greater than 14)
* The family being under-resourced (i.e., family is below the US census poverty line; family is receiving economic or medical government aid; child is receiving reduced fee lunch; or primary caregiver is currently unemployed) or living in an under-resourced community (i.e., majority of households in the family's census block lives under the poverty line).

Exclusion Criteria:

* Current need for acute psychiatric care (e.g., inpatient hospitalization)
* autism spectrum disorder
* psychosis
* other condition(s) related to pronounced cognitive impairment (i.e., marked impairment that precludes completion of questionnaires, verbal communication)
* Wards of the state

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Qualitative interview on acceptability | Posttreatment assessment (week 6)
  Non-numerical identification of narrative textual themes from interviews.
Interpersonal needs questionnaire | Pretreatment (baseline) and week 6
  A 6 question survey assessing thoughts of being a burden on others. Range of possible scores is 6 to 42. Higher scores indicate more severe thoughts of being a burden on others.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Buitron, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided